CLINICAL TRIAL: NCT07370142
Title: Treatment Outcomes of Sphenopalatine Ganglion Pulsed Radiofrequency in Headache Disorders
Brief Title: Sphenopalatine Ganglion Pulsed Radiofrequency Treatment Outcomes
Acronym: SPG-PRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPG-PRF-2025; E2-25-10589 (Other: Ankara Bilkent City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Migraine Disorders, Facial Pain Disorder, Cluster Headache, Trigeminal Neuralgia, Trigeminal Autonomic Cephalalgias
Keywords: Pulsed Radiofrequency; Sphenopalatine Ganglion; Facial Pain; Chronic Headache
MeSH Terms: conditions — Migraine Disorders; Cluster Headache; Trigeminal Neuralgia; Trigeminal Autonomic Cephalalgias; Facial Pain; Headache Disorders

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm interventional study. All participants who meet the inclusion criteria will receive the same intervention (pulsed radiofrequency of the sphenopalatine ganglion). Patients will serve as their own controls, with baseline (pre-procedure) pain scores compared to post-procedure follow-up scores at multiple time points (1 week, 1 month, 3 months, and 6 months)."
Masking Description: No masking is involved in this open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPG Pulsed Radiofrequency Group (Experimental): Patients with refractory chronic headache or facial pain who undergo pulsed radiofrequency (PRF) of the sphenopalatine ganglion under fluoroscopic guidance
  Interventions: Procedure: Pulsed Radiofrequency of the Sphenopalatine Ganglion

INTERVENTIONS:
Procedure: Pulsed Radiofrequency of the Sphenopalatine Ganglion — Fluoroscopy-guided infrazygomatic approach. A 22-gauge, 10-cm RF needle is placed in the pterygopalatine fossa. Pulsed radiofrequency (PRF) is applied at 45V, with 20-ms pulses and 480-ms silent phases. The procedure aims to achieve neuromodulation without thermal tissue damage (local temperature < 42°C).
  Other Names: Pterygopalatine Ganglion Radiofrequency

SUMMARY:
Purpose of the Study: This study aims to evaluate the clinical effectiveness and long-term outcomes of "Sphenopalatine Ganglion (SPG) Pulsed Radiofrequency (PRF)" treatment in patients with chronic headaches and facial pain. The SPG is a major neural junction for craniofacial pain signaling. PRF is a safe, minimally invasive technique that modulates pain transmission without causing thermal damage to the nerve tissue.

Methodology: The study will include at least 30 volunteer patients at the Ankara Bilkent City Hospital Algology Clinic who are unresponsive to medical treatments. Patients will undergo the standard "fluoroscopy-guided infrazygomatic approach." Pain intensity (VAS), quality of life, patient satisfaction, and changes in analgesic consumption will be recorded at baseline and during follow-up visits at 1 week, 1 month, 3 months, and 6 months post-procedure using various clinical parameters.

Expected Benefits and Risks: The research intends to provide evidence regarding the 6-month long-term impact of this intervention on pain scores and patient well-being. Since the study follows routine clinical practices, it poses no additional risks to participants and aims to optimize future treatment strategies.

DETAILED DESCRIPTION:
Study Design and Population This single-center, prospective study involves at least 30 patients diagnosed with chronic headaches and facial pain disorders, including Cluster Headache, Chronic Migraine, Trigeminal Neuralgia, and other Trigeminal Autonomic Cephalalgias (TACs). Participants are selected from patients who have been symptomatic for more than 3 months and are refractory to conventional medical treatments.

Interventional Procedure All procedures are performed in the operating room under fluoroscopic guidance, following the routine clinical practice of the Algology Department:

Positioning: Patients are placed in the supine position. A lateral fluoroscopic view of the face is obtained, ensuring the mandibular rami are superimposed.

Needle Placement: A 22-gauge, 10-cm curved radiofrequency (RF) needle with a 5-mm active tip is advanced via the infrazygomatic approach toward the pterigopalatine fossa.

Confirmation: Proper needle tip positioning is confirmed by intermittent anteroposterior (AP) imaging and sensory stimulation (50 Hz, <0.5 V), aimed at eliciting paresthesia in the maxillary nerve distribution.

Application: Once the position is verified and intravascular entry is ruled out, Pulsed Radiofrequency (PRF) is applied at 45 V with 20-ms bursts and 480-ms silent phases, maintaining a local temperature below 42°C to prevent thermal tissue damage.

Outcome Measures and Follow-up The study evaluates the efficacy and safety of the procedure over a 6-month period. Data collection is performed at baseline (pre-procedure) and post-procedure at 1 week, 1 month, 3 months, and 6 months.

The primary and secondary parameters include:

Pain Intensity: Measured using the Visual Analog Scale (VAS) and Numerical Rating Scale (NRS).

Clinical Efficacy: Assessed via the Global Perceived Effect (GPE) scale (7-point scale ranging from "very much improved" to "very much worse").

Patient Satisfaction: Measured using a 5-point Likert Scale.

Medication Consumption: Changes in analgesic and prophylactic drug use (4-point Likert scale: stopped,increased, stable, or decreased).

Safety Profile: Monitoring for any procedure-related side effects or complications during and after the PRF application.

Statistical Analysis Data will be analyzed using SPSS 25.0. Quantitative data will be tested for normality using Kolmogorov-Smirnov/Shapiro-Wilk tests. Repeated Measures ANOVA or Friedman tests will be utilized to compare longitudinal data across the five time points (baseline to 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older (no upper age limit)
* Patients diagnosed with refractory chronic headache (including cluster headache, migraine, paroxysmal hemicrania, hemicrania continua, SUNCT, or SUNA) or chronic orofacial pain / trigeminal neuralgia
* Pain duration of at least 3 months
* Pain intensity score (VAS or NRS) > 3 out of 10
* Patients unresponsive to conservative medical treatments
* Patients scheduled for sphenopalatine ganglion (SPG) pulsed radiofrequency (PRF) treatment as part of routine clinical care
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Systemic infection or local skin infection at the needle insertion site
* Known coagulopathy or bleeding disorders
* Presence of a cardiac pacemaker or implantable cardioverter-defibrillator (ICD)
* Presence of an intracranial mass or significant anatomical distortion in the pterygopalatine fossa region
* Previous surgical intervention involving the sphenopalatine ganglion
* Pregnancy or breastfeeding
* Severe psychiatric or cognitive disorders preventing reliable pain assessment or follow-up
* Hemodynamic instability
* Refusal to participate in the study or undergo the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain Intensity Reduction Using the Visual Analog Scale (VAS) Following Sphenopalatine Ganglion Pulsed Radiofrequency | "Baseline, 1 week, 3 months, and 6 months post-procedure
  "The Visual Analog Scale (VAS) is a validated measurement tool used to assess pain intensity. It consists of a 10-cm (100-mm) horizontal line anchored by two verbal descriptors: 'no pain' (score 0) and 'the worst imaginable pain' (score 10). Patients are asked to mark the point on the line that represents their current pain level. Lower scores indicate a reduction in pain intensity and an improvement in the patient's clinical status."
Change in Pain Intensity via Visual Analog Scale (VAS) | Baseline, 1 week, 3 months, and 6 months post-procedure.
  A scale ranging from 0 (no pain) to 10 (worst imaginable pain). The goal is to measure the reduction in pain scores compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nevcihan ŞAHUTOĞLU BAL, MD, Principal Investigator — Ankara Bilkent City Hospital, Department of Algology
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To ensure participant privacy and confidentiality, individual participant data will not be shared with outside researchers.